CLINICAL TRIAL: NCT07384689
Title: MiAMII Study - Microdialysis Acquired SaMpling of Ischemia, Inflammation and Antibiotics Locally in Amputation Stump: A Comparative Study in Diabetic and Non-Diabetic Patients Undergoing Non-Traumatic Transfemoral Amputation
Brief Title: Microenvironment in Patients Undergoing Non-traumatic Amputation
Acronym: MiAMII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Rehne Lessmann Hansen, Senior registrar at the department of Orthopaedic Surgery, Amputation and infections unit, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115908
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lower Limb Amputation Above Knee
MeSH Terms: interventions — Silver Sulfadiazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ciNPWT (Active Comparator)
  Interventions: Device: ciNPWT
- SSD (Active Comparator)
  Interventions: Other: SSD

INTERVENTIONS:
Device: ciNPWT — Closed incision negative pressure wound therapy
  Arms: ciNPWT
Other: SSD — Standard stump dressing
  Arms: SSD

SUMMARY:
The microenvironment of the amputation stump in patients undergoing non-traumatic transfemoral amputation will be investigated with a combination of microdialysis and tissue sampling.

ELIGIBILITY:
Inclusion criteria

* 18 years or older
* Cognitive ability to provide informed consent
* Scheduled for transfemoral amputation at Aarhus University Hospital

Exclusion criteria

* Non-vascular indication of amputation
* Already amputated on the contralateral leg
* Insufficient flap perfusion
* Allergic or sensitivity to silver or acrylic adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Ischemia | Within 72 hours postoperatively
  Concentration of ischemic metabolites: Glucose, Lactate, Pyruvate and Glycerol

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark